CLINICAL TRIAL: NCT02005952
Title: Effectiveness of Two Methods for Quality Control in Primary Care Spirometry
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: 09/078/992
Record Dates: First submitted 2013-11-26; First posted 2013-12-09 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2009-05

CONDITIONS: Spirometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Spirometry, quality control, Pulmonary Function Laboratory: Performing spirometry, with control over the quality of the same, made from the pulmonary function laboratory of the Hospital de la Santa Creu i Sant Pau.
- Spirometry, quality control, software: Performing spirometry, with the support of software self-management quality of spirometry maneuvers incorporated therein
- Spirometry, quality control, control group: Performing spirometry in the way that is currently working in primary care (control group without any support).

SUMMARY:
Still not well resolved access, execution and interpretation of spirometry in primary care medicine. This seriously affects the quality of care of chronic respiratory diseases.

OBJECTIVE: To compare the effectiveness of two methods for quality control in performing spirometry in primary care teams (EAP) participating in the "Healthcare Process Chronic Obstructive Pulmonary Disease (COPD )" (multidisciplinary program between primary care medicine and hospital for improved care COPD).

METHODS: Randomized controlled trial of clusters of EAP participants ( n = 17 ). The quality control of spirometry in each EAP randomize into three branches:

1. Supervision from the pulmonary function laboratory of the Hospital ; computer.
2. Program incorporated into automated spirometer.
3. Spirometric usual practice (control group without any support on the quality ). Spirometry EAP participants include year follow-up study . All sites use the same model spirometer and have received the same previous training . In a 2nd phase results implementing the most effective method shown in the 1st phase was studied.

EXPECTED RESULTS : The method for quality control more effective to obtain and maintain the quality spirometry.

POTENTIAL IMPACT EXPECTED : performing spirometry quality in the EAP , improve early detection (secondary prevention ) , the diagnosis of the severity and developmental control of COPD.

ELIGIBILITY:
Inclusion Criteria:

* All patients seen in the participating primary care, requiring spirometry for both the diagnosis and control of any disease will be included.

Exclusion Criteria:

* Patients under 15 years

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients requiring spirometry performing a diagnostic or tracking control for respiratory disease
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2010-02; Primary Completion 2011-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Effectiveness of two methods for quality control in primary care spirometry | Basal

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Giner, MSc, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau